CLINICAL TRIAL: NCT00975637
Title: A Randomized, Double-blind, Placebo-controlled, Multiple-dose Study to Evaluate the Safety, Tolerability, and Efficacy of AMG 827 in Subjects With Psoriasis
Brief Title: Study to Evaluate the Safety, Tolerability, and Efficacy of AMG 827 in Subjects With Psoriasis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bausch Health Americas, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 20090062
Record Dates: First submitted 2009-09-10; First posted 2009-09-11 (Estimated); Results first posted 2016-12-30 (Estimated); Last update posted 2019-06-26 (Actual); Status verified 2019-06

CONDITIONS: Psoriasis
MeSH Terms: conditions — Psoriasis | interventions — brodalumab

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (5):
- 140 mg SC (Experimental): 140 mg SC
  Interventions: Drug: 140 mg SC
- 70 mg SC (Experimental): 70 mg SC
  Interventions: Drug: 70 mg SC
- 280 mg SC (Experimental): 280 mg SC
  Interventions: Drug: 280 mg SC
- 210 mg SC (Placebo Comparator): 210 mg SC
  Interventions: Drug: 210 mg SC
- Placebo (Experimental): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: 70 mg SC — 70 mg SC
  Other Names: AMG 827
  Arms: 70 mg SC
Drug: 210 mg SC — 210 mg SC
  Other Names: AMG 827
  Arms: 210 mg SC
Drug: 140 mg SC — 140 mg SC
  Other Names: AMG 827
  Arms: 140 mg SC
Drug: 280 mg SC — 280 mg SC
  Other Names: AMG 827
  Arms: 280 mg SC
Drug: Placebo — Placebo SC
  Arms: Placebo

SUMMARY:
The study evaluated the efficacy of AMG 827 compared with placebo as measured by the percent of improvement in PASI score at week 12.

DETAILED DESCRIPTION:
The study evaluated the efficacy of AMG 827 compared with placebo as measured by the percent of improvement in PASI score at week 12. Subjects were randomized ina 1:1:1:1:1 ratio. Subjects randomized to receive AMG 827 received 70, 140, or 210 mg at day 1 and weeks 4 and 8.

ELIGIBILITY:
Inclusion Criteria:

* Subject has had stable moderate to severe plaque psoriasis for at least 6 months
* Subject has received at least one previous phototherapy or systemic psoriasis therapy or has been a candidate to receive phototherapy or systemic psoriasis therapy in the opinion of the investigator.
* Subject has involved BSA ≥ 10% and PASI ≥ 12 at screening and at baseline.

Exclusion Criteria:

* Subject diagnosed with erythrodermic psoriasis, pustular psoriasis, medication-induced, or medication-exacerbated psoriasis.
* Evidence of skin conditions at the time of the screening visit (eg, eczema, guttate psoriasis) that would interfere with evaluations of the effect of IP on psoriasis.
* Subject has any active CTCAE grade 2 or higher infection
* Subject has a significant concurrent medical condition or laboratory abnormalities, as defined in the study protocol.
* Subject has used the following therapies within 14 days of the first dose: UVB therapy or topical psoriasis therapies other than Class I or II topical steroids
* Subject has used the following therapies within 28 days of the first dose: Class I or II topical steroids, UVA therapy (with or without psoralen), or systemic psoriasis therapies
* Subject has used the following therapies within 3 months of the first dose: adalimumab, alefacept, etanercept, infliximab, certolizumab, or live vaccines
* Subject has used an anti-IL12/IL23 inhibitor within 6 months of the first dose
* Subject has previously used an anti-IL17 biologic therapy, efalizumab, or rituximab

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 198 (Actual)
Dates: Start 2009-12; Primary Completion 2010-07 (Actual); Study Completion 2010-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Gordon KB, Kimball AB, Chau D, Viswanathan HN, Li J, Revicki DA, Kricorian G, Ortmeier BG. Impact of brodalumab treatment on psoriasis symptoms and health-related quality of life: use of a novel patient-reported outcome measure, the Psoriasis Symptom Inventory. Br J Dermatol. 2014 Mar;170(3):705-15. doi: 10.1111/bjd.12636. PMID 24079852
- [Background] Papp KA, Leonardi C, Menter A, Ortonne JP, Krueger JG, Kricorian G, Aras G, Li J, Russell CB, Thompson EH, Baumgartner S. Brodalumab, an anti-interleukin-17-receptor antibody for psoriasis. N Engl J Med. 2012 Mar 29;366(13):1181-9. doi: 10.1056/NEJMoa1109017. PMID 22455412
- [Background] Papp K, Menter A, Strober B, Kricorian G, Thompson EH, Milmont CE, Nirula A, Klekotka P. Efficacy and safety of brodalumab in subpopulations of patients with difficult-to-treat moderate-to-severe plaque psoriasis. J Am Acad Dermatol. 2015 Mar;72(3):436-439.e1. doi: 10.1016/j.jaad.2014.10.026. Epub 2014 Dec 29. PMID 25553889
- [Derived] Gottlieb A, Lebwohl M, Liu C, Israel RJ, Jacobson A. Malignancy Rates in Brodalumab Clinical Studies for Psoriasis. Am J Clin Dermatol. 2020 Jun;21(3):421-430. doi: 10.1007/s40257-020-00512-4. PMID 32207067
- [Derived] Papp K, Leonardi C, Menter A, Thompson EH, Milmont CE, Kricorian G, Nirula A, Klekotka P. Safety and efficacy of brodalumab for psoriasis after 120 weeks of treatment. J Am Acad Dermatol. 2014 Dec;71(6):1183-1190.e3. doi: 10.1016/j.jaad.2014.08.039. Epub 2014 Oct 11. PMID 25313095
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Groups:
- 210 mg: AMG 827: 210 mg SC
- 140 mg: AMG 827: 140 mg SC
- 280 mg: AMG 827: 280 mg SC
- 70 mg: AMG 827: 70 mg SC
Period: Overall Study
Arm/Group | 210 mg | 140 mg | 280 mg | Placebo | 70 mg
Started | 40 | 39 | 42 | 38 | 39
Completed | 37 | 38 | 40 | 32 | 37
Not Completed | 3 | 1 | 2 | 6 | 2

BASELINE CHARACTERISTICS:
Groups:
- Broda 210 mg: AMG 827: 210 mg SC
- Broda 140 mg: AMG 827: 140 mg SC
- Broda 280 mg: AMG 827: 280 mg SC
- Broda 70 mg: AMG 827: 70 mg SC
- Total: Total of all reporting groups
Arm/Group | Broda 210 mg | Broda 140 mg | Broda 280 mg | Placebo | Broda 70 mg | Total
Number analyzed (Participants) | 40 | 39 | 42 | 38 | 39 | 198
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 39 | 38 | 40 | 35 | 38 | 190
  >=65 years | 1 | 1 | 2 | 3 | 1 | 8
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.1 (12.2) | 44.0 (11.7) | 42.3 (12.2) | 41.8 (14.4) | 42.1 (11.1) | 42.6 (11.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 11 | 12 | 16 | 17 | 71
  Male | 25 | 28 | 30 | 22 | 22 | 127
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 1 | 0 | 2 | 1 | 6
  Not Hispanic or Latino | 38 | 38 | 41 | 36 | 38 | 191
  Unknown or Not Reported | 0 | 0 | 1 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Dose-response Efficacy Profile of AMG 827 Compared With Placebo as Measured by the Percent Improvement From Baseline in Psoriasis Area and Severity Index (PASI) Score at Week 12
Description: At screening a subject would need to have a PASI score of equal to or greater than 12, so at week 12 they were assessed to see percentage of change from there baseline PASI score.
Time Frame: Baseline and 12 weeks
Measure: Mean (Standard Deviation); unit: percentage of psoriasis improvement
Arm/Group | Broda 210 mg | Broda 140 mg | Broda 280 mg | Placebo | Broda 70 mg
Number analyzed (Participants) | 40 | 39 | 42 | 38 | 39
percentage of psoriasis improvement | 86.3 (27.6) | 85.9 (22.5) | 76 (32.7) | 16 (27) | 45 (41.7)

2. Secondary Outcome: Change in Percent of Body Surface Area (BSA) Affected by Psoriasis
Description: To evaluate the efficacy of AMG 827 as measured by the following: Body surface area (BSA) involvement at weeks 12. At the baseline of the study the subject would need to have at least a 10% BSA; at week 12 they were again assessed to see what change in percentage of BSA has occurred.
Time Frame: Baseline and Week 12
Measure: Mean (Standard Deviation); unit: percentage improvement in BSA
Arm/Group | Broda 210 mg | Broda 140 mg | Broda 280 mg | Placebo | Broda 70 mg
Number analyzed (Participants) | 40 | 39 | 42 | 38 | 39
percentage improvement in BSA | 22.1 (15.0) | 21.1 (16.9) | 16.1 (11.4) | 0.9 (9.7) | 9.2 (11.2)

ADVERSE EVENTS:
Arm/Group | Broda 210 mg | Broda 140 mg | Broda 280 mg | Placebo | Broda 70 mg
Serious Adverse Events (participants affected / at risk) | 1/40 | 0/39 | 0/42 | 0/38 | 0/39
Other Adverse Events (participants affected / at risk) | 15/40 | 12/39 | 10/42 | 7/38 | 10/39
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Broda 210 mg (N=40) | Broda 140 mg (N=39) | Broda 280 mg (N=42) | Placebo (N=38) | Broda 70 mg (N=39)
Neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Broda 210 mg (N=40) | Broda 140 mg (N=39) | Broda 280 mg (N=42) | Placebo (N=38) | Broda 70 mg (N=39)
Injection Site Erythema (General disorders) | 3 | 1 | 4 | 1 | 1
Injection Site Pain (General disorders) | 0 | 0 | 1 | 0 | 3
Fatigue (General disorders) | 2 | 2 | 0 | 0 | 1
Injection Site Induration (General disorders) | 1 | 0 | 2 | 0 | 0
Injection Site Swelling (General disorders) | 1 | 1 | 1 | 0 | 0
Injection Site Pruritus (General disorders) | 0 | 1 | 1 | 1 | 0
Injection Site Hematoma (General disorders) | 0 | 0 | 0 | 0 | 1
Injection Site Uticaria (General disorders) | 0 | 0 | 1 | 0 | 0
Injection Site Warmth (General disorders) | 0 | 1 | 0 | 0 | 0
Chills (General disorders) | 0 | 0 | 0 | 1 | 0
Oedema Peripheral (General disorders) | 0 | 0 | 0 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 1 | 1 | 0 | 2
Furuncle (Infections and infestations) | 1 | 1 | 1 | 0 | 0
Bronchitis (Infections and infestations) | 1 | 0 | 0 | 1 | 1
Nasopharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 2
Abscess Limb (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Herpes Zoster (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Oral candidiasis (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Oral Herpes (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Pharnyngitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Sinustitis (Infections and infestations) | 0 | 0 | 1 | 1 | 0
Viral Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Psoriasis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 1 | 0
Acne (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
Mechanical Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Rash Morbilliform (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No